CLINICAL TRIAL: NCT06191367
Title: Effect of Aerobic Exercises Versus Incentive Spirometer Device on Post-covid Pulmonary Fibrosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McCarious Nahad Aziz Abdelshaheed Stephens (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, McCarious Nahad Aziz Abdelshaheed Stephens, Researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CairoU post-covid PF Rehab
Record Dates: First submitted 2023-12-23; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Lung Fibrosis Interstitial; Post-COVID-19 Syndrome
MeSH Terms: conditions — Pulmonary Fibrosis; Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (experimental) Aerobic Exercises and Traditional Chest Physiotherapy. (Experimental): It was consisted of fifteen patients with positive covid-19 test from at least a month before trial. They received aerobic exercise techniques which consist of 3 levels of activity exercises and traditional program of chest physiotherapy. (Five times per week for two months).
  Interventions: Other: Aerobic Exercises; Other: Traditional Chest Physiotherapy
- Group II (experimental)Incentive Spirometer Device and Traditional Chest Physiotherapy. (Experimental): It was consisted of fifteen patients with positive covid-19 test from at least a month before trial. They received incentive spirometer training techniques and traditional program of chest physiotherapy. (Five times per week for two months).
  Interventions: Device: Incentive Spirometer Device; Other: Traditional Chest Physiotherapy
- Group III (control) will receive Traditional Chest Physiotherapy only. (Active Comparator): As a control group it was consisted of fifteen patients with positive covid-19 test from at least a month before trial. They received traditional program of chest physiotherapy only. (Five times per week for two months).
  for example: - Breathing Exercises. - Postural Drainage. - Percussion. - Coughing - Vibration.
  Interventions: Other: Traditional Chest Physiotherapy

INTERVENTIONS:
Other: Aerobic Exercises — Aerobic Exercises
  Arms: Group I (experimental) Aerobic Exercises and Traditional Chest Physiotherapy.
Device: Incentive Spirometer Device — is a handheld medical device used to help patients improve the functioning of their lungs. By training patients to take slow and deep breaths, this simplified spirometer facilitates lung expansion and strengthening. Patients inhale through a mouthpiece, which causes a piston inside the device to rise. This visual feedback helps them monitor their inspiratory effort. Incentive spirometers are commonly used after surgery or other illnesses to prevent pulmonary complications.
  Arms: Group II (experimental)Incentive Spirometer Device and Traditional Chest Physiotherapy.
Other: Traditional Chest Physiotherapy — 1. Breathing exercise.
  2. Postural drainage.
  3. Percussion.
  4. Coughing.
  5. Vibration.

SUMMARY:
the aim of this study will be to investigate the effect of aerobic exercises vs incentive spirometer device on post-covid patients with residual lung diseases.

DETAILED DESCRIPTION:
To our knowledge, there have been no enough studies that investigated the effect of aerobic exercise and incentive spirometer in pulmonary rehabilitation on post-covid syndrome patients.

Therefore, this study may open up ways to other researchers to investigate and build up on this effect if present and address such an important issue.

The finding of this proposed work may help patients with post-covid syndrome and complain of lung diseases by addressing their complains of symptoms like chest pain, dyspnea, and cough and provide a possible solution to enhance their quality of life and increase their participation in daily life activities.

Patients of post-covid syndrome with residual lung problems will be recruited after approval of ethical committee of the faculty of physical therapy, Cairo university. All participants will sign a written informed consent form.

The subjects will be randomly assigned into one of three groups:

* Group I (experimental) will receive aerobic exercises program and traditional chest physiotherapy.
* Group II (experimental) will receive incentive spirometer device treatment and traditional chest physiotherapy.
* Group III (control) will receive traditional chest physiotherapy only. The measures will be taken before and after treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamic stable (MAP not less than 60mmHg, systolic pressure >80mmHg and diastolic pressure not <60mmHg)
* Age from 40 to 85 years.
* Both sexes.
* All patients were positive covid-19 infected patients and passed at least 4 weeks after confirmation.
* All patients suffer from respiratory complications.
* All patients included are actively breathing.
* All patients included are fully aware and conscious.

Exclusion Criteria:

* Hemodynamic Instability.
* Severe Head Injury.
* Increased intracranial pressure.
* Anemic Hb<8.
* Active Smoking.
* Severe Bronchospasm.
* Low BP (systole <80, diastole <60).
* Subcutaneous Emphysema.
* Rip Fractures.
* Untreated Pneumothorax.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function tests (PFTs). | Before and After the treatment program. "8 weeks"
  to measure the lungs' capacities and volumes like: FVC, FEV1, and PEF.
Peripheral oxygen saturation level (SpO2). | Before and After the treatment program. "8 weeks"
  measures the amount of oxygen carried in the blood stream in peripheral limbs.
Six minutes' walk distance test (6MWD). | Before and After the treatment program. "8 weeks"
  measures the aerobic capacity of the lungs by testing the maximum distance the subject can walk in a 6 minutes time.
Heart rate measurements. (HR). | through all the treatment procedures. "8 weeks"
  it measures the number of heart bumps in a minute in order to deliver blood to all of the body during Rest and Activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Elgendy, Doctoral, Principal Investigator — Physiotherapy Faculty, Cairo University.
Locations (1):
- Physiotherapy department Police Academy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Undecided